CLINICAL TRIAL: NCT03644212
Title: Vitamin D Increases Serum Levels of the Soluble Receptor for Advanced Glycation End Products in Women With PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/07/XA03
Record Dates: First submitted 2013-05-04; First posted 2018-08-23 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Polycystic Ovary Syndrome; Vitamin D Deficiency
Keywords: Polycystic Ovary Syndrome; Vitamin D; Anti Mullerian Hormone; Soluble receptor for Advanced Glycation End Products
MeSH Terms: conditions — Polycystic Ovary Syndrome; Vitamin D Deficiency | interventions — Cholecalciferol; Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D treatment (Active Comparator): Sixty-three vitamin D deficient women (16 with PCOS and 47 without PCOS) were supplemented with 50.000 IU of oral vitamin D3, once weekly for 8 weeks. Serum 25-hydroxyvitamin D (25OH-D), sRAGE and AMH levels were checked before and after treatment.
  Interventions: Drug: Vitamin D3
- Non treated (No Intervention): Sixteen vitamin D deficient women (6 with PCOS and 10 without PCOS) were not supplemented vitamin D3. Serum 25-hydroxyvitamin D (25OH-D), sRAGE and AMH levels were checked before and after treatment.

INTERVENTIONS:
Drug: Vitamin D3 — Sixty-three vitamin D deficient women (16 with PCOS and 47 without PCOS) were supplemented with 50.000 IU of oral vitamin D3, once weekly for 8 weeks. Serum 25-hydroxyvitamin D (25OH-D), sRAGE and AMH levels were checked before and after treatment.
  Other Names: Vitamin
  Arms: Vitamin D treatment

SUMMARY:
The purpose of this study is to investigate the mechanism that explain the beneficial clinical effect of vitamin D treatment in women with PCOS.

DETAILED DESCRIPTION:
Seventy-nine women with (n=22) or without (control; n=57) PCOS who were diagnosed with vitamin D deficiency were enrolled. Sixty-three women were treated with oral vit D3 for 8 weeks (16 with PCOS and 47 controls) and 16 women were not treated (6 with PCOS and 10 controls). Serum 25 hydroxy-vitamin D (25 OH-D), sRAGE, and AMH concentrations were measured at baseline and after vit D3 supplementation in the treated group, and 8 weeks apart in the non-treated group. Paired t-test, Wilcoxon signed-rank test, and Pearson correlation were used as appropriate.

Main outcome measure: Changes in AMH concentrations following vit D3 replacement.

ELIGIBILITY:
Inclusion Criteria:

* Vitamin D deficient premenopausal women

Exclusion Criteria:

* Pregnant women
* Women during their postpartum period
* Breastfeeding women
* Women taking any kind of exogenous hormones
* Women receiving any form of oral vitamin D replacement

Ages: 16 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Irani, MD, Study Director — Maimonides Medical Center, Brooklyn, NY, USA; Zaher Merhi, MD, Principal Investigator — University of Vermont College of Medicine, Burlington, VT, USA
Locations (1):
- Maimonides Medical Center, OBGYN clinic, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D Treatment | Non Treated
Started | 63 | 16
Completed | 63 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D Treatment | Non Treated | Total
Number analyzed (Participants) | 63 | 16 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 16 | 79
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 16 | 79
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 16 | 79

OUTCOME MEASURES:

1. Primary Outcome: AMH Levels in Women With PCOS
Description: AMH measured by serum analysis
Time Frame: 8 weeks after completing vitamin D treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D Treatment | Non Treated
Number analyzed (Participants) | 63 | 16
ng/mL | 1.4 (0.55) | 0 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the 8 weeks of the study.
Arm/Group | Vitamin D Treatment | Non Treated
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/16
Other Adverse Events (participants affected / at risk) | 0/63 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes